CLINICAL TRIAL: NCT06799520
Title: A Phase 1 Open-label Trial to Evaluate the Safety, Tolerability, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of Subcutaneous VIS171 in Participants With Autoimmune Disease(s)
Brief Title: A Phase 1 Trial to Evaluate the Safety, Tolerability, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of VIS171 in Participants With Autoimmune Disease(s)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIS171-103; 2024-518976-30 (Other: EU Trial Number)
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus (SLE); Alopecia Areata (AA); Immune-mediated Focal Segmental Glomerulosclerosis (FSGS)
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VIS171 (Experimental): Participants will receive VIS171 dose via SC injection, from Week 1 to Week 21.
  Interventions: Drug: VIS171

INTERVENTIONS:
Drug: VIS171 — VIS171 will be administered as a SC injection.

SUMMARY:
The purpose of this trial is to measure safety and tolerability of subcutaneous (SC) VIS171 in combination with standard of care in participants with autoimmune disease(s). The total duration of the clinical trial for each participant will be up to approximately 9 to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Estimated glomerular filtration rate (eGFR) >30 milliliters/minute/1.73 square meters (mL/min/1.73 m^2) at the screening visit.

   For SLE participants:
2. Participant has a confirmed diagnosis of SLE according to European League Against Rheumatism/American College of Rheumatology SLE classification criteria ≥ 24 weeks prior to signing the informed consent form (ICF).

   For AA participants:
3. Current scalp involvement between 25% and 95%, inclusive (Severity of Alopecia Tool [SALT] score between 25 and 95, inclusive), at screening.
4. Current episode of AA is of duration > 24 weeks (without evidence of spontaneous terminal hair regrowth at the time of screening and first treatment, i.e., no more than 10% regrowth), but ≤ 5 years from onset of current episode of severe scalp hair loss.

   For FSGS participants:
5. Prior biopsy (no time limit) showing histologic minimal change disease (MCD), FSGS, or MCD/FSGS spectrum.
6. History of at least one prior episode of nephrotic syndrome, defined as 24-hour urine protein > 3.5 grams per day (g/day) and serum albumin < 3.5 grams per deciliter (g/dL).
7. History of steroid responsive nephrotic syndrome, including participants who achieved complete remission, partial remission, had a course of steroid dependent nephrotic syndrome or relapsing nephrotic syndrome (all defined as per the managing physician at the time of the episode).

Exclusion Criteria:

1. Receipt of high-dose corticosteroid therapy within 4 weeks prior to screening as either (a) intravenous (IV) pulse corticosteroid therapy or (b) daily oral corticosteroid therapy of ≥ 1 milligrams per kilogram (mg/kg) or up to 40 milligrams per day (mg/day) prednisone (or equivalent).
2. Receipt of blood products within 6 months prior to screening.
3. Previous exposure to VIS171 or any other drug targeting interleukins (IL)-2 or the IL-2 receptor or T regulatory cells.
4. History of or current diagnosis of catastrophic or severe anti-phospholipid syndrome (APS) within 1 year prior to signing ICF. SLE participants with APS adequately controlled by anticoagulant are eligible. SLE participants who are found to be triple positive for anti-phospholipid antibodies at screening (without clinical APS) will be excluded unless they are on stable anti-thrombotic therapy.
5. Known primary immunodeficiency disorder.
6. Participant has a history of Class V lupus nephritis.
7. Receipt of anifrolumab, tumor necrosis factor-alpha monoclonal antibodies ([TNF]-α mAb), immunoglobulins (IV/SC) plasmapheresis, or any other immunosuppressants (calcineurin inhibitors, Janus kinase [JAK] inhibitors or other kinase inhibitors), other than hydroxychloroquine, mycophenolic acid (MPA)/mycophenolate mofetil (MMF) and corticosteroids, within 6 months prior to screening.
8. Participant has concomitant hair loss of another form, including but not limited to traction alopecia, central centrifugal cicatricial alopecia, lichen planopilaris, frontal fibrosing alopecia, or androgenetic alopecia.
9. Participant has received (1) Within 12 weeks prior to Day 1: Systemic therapies (oral or injection), such as corticosteroids, JAK inhibitors, methotrexate, calcineurin inhibitors, oral minoxidil, low-dose IL-2 and topical immunotherapies such as psoralen plus UVA (PUVA) , diphenylcyclopropenone (DPCP), dinitrochlorobenzene (DNCB), intralesional steroids or (2) Within 4 weeks prior to Day 1: Other topical therapies, such as topical minoxidil, clobetasol etc. These therapies will also not be allowed during this trial.
10. Steroid resistant nephrotic syndrome defined as absence of history of at least 1 episode of complete or partial remission following at least 12 weeks of full dose corticosteroid therapy.
11. Receipt of anifrolumab, TNF-α mAb, immunoglobulins (IV/SC) plasmapheresis, or any other immunosuppressants (JAK inhibitors or other kinase inhibitors).

Note: Other protocol-specified Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) Graded by Severity | From first dose of the study drug up to end of the study (up to Week 45)

SECONDARY OUTCOMES:
Change from Baseline in Absolute Number of Regulatory T (Treg) Cells, Total T Helper Cells, Cytotoxic T Cells, and Natural Killer Cells in Blood | From baseline up to Week 21
Percent Change from Baseline in Treg Cells/CD4+ Cells, Total T Helper Cells, Cytotoxic T Cells, and Natural Killer Cells in Blood | From baseline up to Week 21
Serum Concentration of VIS171 Over Time | Up to Week 21
Number of Participants with Confirmed Positive or Negative Anti-drug Antibody (ADA) Titers | Up to Week 21

CONTACTS AND LOCATIONS:
Locations (6):
- Visterra Investigational Site, Sofia, Bulgaria
- Visterra Investigational Site, Chisinau, Moldova
- Romania (2):
  - Visterra Investigational Site, Bucharest
  - Visterra Investigational Site, Cluj-Napoca
- Spain (2):
  - Visterra Investigational Site, Barcelona
  - Visterra Investigational Site, Granada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets,or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com